CLINICAL TRIAL: NCT00327886
Title: A Retrospective Review of Postoperative Management of Cyanosis Following Bidirectional Glenn Operation
Brief Title: Managing Cyanosis Following Bidirectional Glenn Operation
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 06-029
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Congenital Disorders
Keywords: pediatric; Glenn operation; Cyanosis
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Cyanosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this retrospective study is to review the postoperative medical management of infants who underwent bidirectional Glenn operation from January 1, 2003 to December 31, 2005 who were significantly cyanotic.

DETAILED DESCRIPTION:
Infants following bidirectional Glenn operation are at times significantly cyanotic. The medical management of significant postoperative cyanosis has changed with the advent of nitric oxide, sildenafil and bosentan. The purpose of this retrospective study is to review the postoperative medical management of infants who underwent bidirectional Glenn operation from Jan 1, 2003 to Dec 31, 2005 who were significantly cyanotic.

Summary of Procedures This is a retrospective study, therefore, the only procedure will be a chart review. I estimate the number of patients to be around 150, however, request permission to review the patient population in order to provide exact numbers. We request permission to review hospital charts from the time of bidirectional Glenn operation and the last clinic note within the dates Jan 1, 2003 to Dec 31, 2005.

We will assign each chart a unique study number and collect data of:

date of follow-up oxygen saturation during stay time since discharge 02 saturation at home home medications when discontinue medications

ELIGIBILITY:
Inclusion Criteria:

* Infants
* Bidirectional Glenn operation between 1/1/03-12/31/05
* Significant Cyanosis

Exclusion Criteria:

* Those who do not meet inclusion criteria.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2006-02; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Simsic, MD, Principal Investigator — Sibley Heart Center Cardiology, Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States